CLINICAL TRIAL: NCT02032303
Title: Assessment of Coronary Flow Reserve by Doppler Flow WIre in Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention: Differences Between the Loading Dose of Prasugrel and Ticagrelor .
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Massimo Mancone, PhD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Ticagrelor - Prasugrel
Record Dates: First submitted 2013-12-18; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Acute Coronary Syndrome; Non ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Angina, Unstable | interventions — Percutaneous Coronary Intervention

ARMS (2):
- Ticagrelor (Active Comparator): Patient randomized to Ticagrelor
  Interventions: Procedure: Assessment of coronary flow reserve; Procedure: Percutaneous Coronary Intervention; Drug: Ticagrelor loading
- Prasugrel (Active Comparator): Patient randomized to Prasugrel
  Interventions: Procedure: Assessment of coronary flow reserve; Procedure: Percutaneous Coronary Intervention; Drug: Prasugrel loading

INTERVENTIONS:
Procedure: Assessment of coronary flow reserve
Procedure: Percutaneous Coronary Intervention
Drug: Ticagrelor loading
  Arms: Ticagrelor
Drug: Prasugrel loading
  Arms: Prasugrel

SUMMARY:
Study design Investigators aim to perform a prospective, single-center, investigator-initiated, randomized study to compare the Adenosine-induced coronary vasodilatation after the loading dose of Ticagrelor either Prasugrel during the Percutaneous Coronary Intervention. Patients with acute coronary syndrome undergoing Percutaneous Coronary Intervention will be enrolled in the study and will be randomized, in a 1:1 ratio, to receive a loading dose of Ticagrelor (180 mg) or Prasugrel (60 mg). In patients with non-ST elevation myocardial infarction these drugs will be administered only when the coronary anatomy will be known, to avoid bleeding due to prasugrel, in patients suitable for coronary artery bypass grafting as recommended by European Society of Cardiology guidelines (Class IB) (10). In patients with ST elevation myocardial infarction, instead, prasugrel and ticagrelor will be administrated before the procedure, according to the European Society of Cardiology guidelines (Class IB) (11). Coronary Flow Reserve will be recorded by intracoronary Doppler Flow Wire before the stent implantation and after the procedure at baseline and 2-minute later adenosine intravenous administration at incremental doses of 50, 80, 110 and 140 ug/Kg/min with 2 minutes interval between infusions.

Coronary Flow Reserve is the ability of the myocardium to increase blood flow in response to maximal exercise. Doppler Flow Wire allows to measure this increase expressing it as a ratio between maximal vasodilation and flow at rest. Coronary Flow Reserve is routinely measured in patients with acute coronary syndrome, without an increased risk of adverse events for patients neither adjunctive costs for the National Health System.

Furthermore, Plasma concentrations of Ticagrelor and its main metabolite (AR-C124910XX) will be measured in venous blood collected at the end of the procedure. . In patients requiring a second Percutaneous Coronary Intervention, for example for multivessel disease, all these measures will be repeated in the same manner.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with acute coronary syndrome undergoing Percutaneous Coronary Intervention with stent implantation;

  * Patients ≥ 18 and ≤ 75 years old.
  * Signed informed consent;

Exclusion Criteria:

* • Patients with stable angina;

  * prior myocardial infarction;
  * prior revascularization (Percutaneous Coronary Intervention or coronary artery bypass grafting);
  * Ticagrelor contraindications (history of intracranial hemorrhage, active pathological bleeding, severe hepatic impairment);
  * Prasugrel contraindications (patients weighing less than 60 kg, patients who had previous stroke or transient ischemic attack, patients aged more than 75 years old);
  * major periprocedural complications;
  * suboptimal Percutaneous Coronary Intervention result (residual stenosis > 20%);
  * glomerular filtration rate < 30 ml/min or requiring haemodialysis;
  * Non-sinus rhythm;
  * severe chronic obstructive pulmonary disease;
  * requirement for oral anticoagulant;
  * risk of bleeding or bradycardic events;
  * ejection fraction < 45%;
  * Cardiogenic shock;
  * Severe left ventricular hypertrophy;
  * severe valvular disease;
  * diffuse coronary atherosclerosis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
assessment of coronary flow reserve | 2 hours after the loading dose

CONTACTS AND LOCATIONS:
Locations (1):
- Massimo Mancone, Rome, Rome, Italy